CLINICAL TRIAL: NCT02704221
Title: Enhancing the Outcomes of a Behavioral Parent Training Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christina Studts (Other)
Collaborators: University of Vermont (Other)
Responsible Party: Sponsor-Investigator, Christina Studts, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 15-0291-P6H
Record Dates: First submitted 2016-03-04; First posted 2016-03-09 (Estimated); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Disruptive Behavior Disorder; Parenting
MeSH Terms: conditions — Attention Deficit and Disruptive Behavior Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral Parent Training (BPT) (Active Comparator): The control group will include 10 participants who will 1) wear Fitbit activity trackers daily for 12 weeks and 2) attend 12 weekly BPT training sessions.
  Interventions: Behavioral: Fitbit activity tracker; Behavioral: BPT training sessions
- BPT + Contingency Management (BPT+CM) (Experimental): The experimental group will include 10 participants who will 1) wear Fitbit activity trackers daily for 12 weeks, 2) attend 12 weekly BPT training sessions, and 3) receive monetary rewards for achieving weekly step-count goals.
  Interventions: Behavioral: Fitbit activity tracker; Behavioral: Monetary rewards; Behavioral: BPT training sessions

INTERVENTIONS:
Behavioral: Fitbit activity tracker — Wear a Fitbit daily for 12 weeks and meet with a research assistant once per week to download data
Behavioral: Monetary rewards — Set weekly step-count goals based on the previous week's performance and receive monetary rewards for meeting the goals. The schedule of rewards increases as step-count goals increase.
  Arms: BPT + Contingency Management (BPT+CM)
Behavioral: BPT training sessions — Complete 12 BPT training sessions delivered by supervised clinical child psychology doctoral students, with each session lasting approximately 60 minutes. The BPT is based upon the existing, evidence-based Everyday Parenting intervention.

SUMMARY:
This study is a feasibility trial, testing the hypothesis that among sedentary mothers of behaviorally at-risk preschool-aged children, those who receive behavioral parent training (BPT) programs and concurrently increase their physical activity levels will demonstrate improved parenting and child behavior outcomes compared to those who receive BPT but remain sedentary.

DETAILED DESCRIPTION:
The investigators will randomly assign 20 participants to two groups: behavioral parent training plus contingency management to increase steps (BPT+CM) or behavioral parent training alone (BPT). Contingency management procedures will involve monetary rewards for meeting weekly step-count goals.

The specific aims of the proposed project are to: 1) assess the feasibility of the study design and procedures, 2) assess the acceptability of the BPT+CM condition to participants, and 3) determine whether a signal of an effect of increased physical activity exists (via preliminary comparisons of measures of fatigue, perceived energy, parenting behaviors, parenting sense of competence, parenting stress, and child behavior ratings between participants in the two conditions).

This innovative pilot study will prepare us for a fully powered trial to test the efficacy of this approach.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 18 years or older
* Custodial caregiver of a child aged 2-5 years who lives full-time in the caregiver's home
* Reports that her child has behavioral problems
* Never or rarely engages in regular physical activity
* Able to understand, speak, and read English

Exclusion Criteria:

* The child has been diagnosed with a severe developmental condition (e.g., extreme developmental delay, severe autism, debilitating neurological conditions)
* Participant reports a condition that may contraindicate physical activity (e.g., asthma)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-03-01; Primary Completion 2017-10-01 (Actual); Study Completion 2018-09-13 (Actual)

PRIMARY OUTCOMES:
Proportion of participants who complete study procedures within study timeframe | 14 months

SECONDARY OUTCOMES:
Time required per participant to complete all instruments | 14 months
Participant satisfaction of both control and experimental arms | 1 week after completion of final BPT session
Step counts | end of 2-week screening period, and once per week for 12 weeks
2-minute step test | baseline and 1 week after completion of final BPT session
Parenting behaviors | baseline and 1 week after completion of final BPT session
  Parenting Young Children instrument
Child behaviors | baseline and 1 week after completion of final BPT session
  Child Behavior Checklist/1.5-5 instrument
Parenting stress | baseline and 1 week after completion of final BPT session
  Parenting Stress Index/Short Form instrument
Parenting sense of competence | baseline and 1 week after completion of final BPT session
  Parenting Sense of Competence Scale
Parent depression | baseline and 1 week after completion of final BPT session
  Beck Depression Inventory-II
Self-reported physical activity level | baseline and 1 week after completion of final BPT session
  Godin Leisure-Time Exercise Questionnaire
Visual Analog Scale-Fatigue | baseline and 1 week after completion of final BPT session

CONTACTS AND LOCATIONS:
Overall Officials: Christina Studts, PhD, LCSW, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky General Pediatrics Clinic, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No